CLINICAL TRIAL: NCT01741766
Title: The Effects of 8 Weeks of Stretching Training on Arterial Stiffness, Wave Reflection, Endothelial Function and Cardiac Autonomic Control.
Brief Title: The Effects of Stretching Training on Arterial Function and Autonomic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC2010.5615
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Pre-hypertension; Hypertension
Keywords: prehypertension; hypertension; obesity; stretching; arterial function; arterial stiffness; pulse wave velocity; autonomic function; endothelial function
MeSH Terms: conditions — Obesity; Prehypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stretching Training (Experimental): Whole body stretching exercises 3 times per wk for 8 weeks
  Interventions: Other: Stretching Training
- Control (No Intervention): This arm involves not making any change to the subject's lifestyle at the moment of the start of the intervention and for 8 wk.

INTERVENTIONS:
Other: Stretching Training — The stretching training intervention consists of 38 whole-body stretching exercises, 3 times per week for 8 wk. Each stretch will be held in place for 30 seconds, with a 15 seconds of rest in between stretches.
  Arms: Stretching Training

SUMMARY:
Hypertension is a major risk factor for cardiovascular disease. Hypertension and abdominal obesity are associated with dysfunction of the main mechanisms of cardiovascular regulation, the autonomic nervous system and the vascular endothelium. Increased sympathetic activity and endothelial dysfunction are associated with increased arterial stiffness, which is an independent risk factor for the development of hypertension and other cardiovascular diseases. The recommended intervention for controlling BP in pre- and stage 1- hypertensive individuals is lifestyle modifications such as exercise, and not drug therapy.Although aerobic and resistance exercise has been shown to be beneficial for the cardiovascular system, special populations such as the elderly and obese may have physical and/or musculoskeletal limitations which may limit their participation in these exercise modalities.

Stretching is a form of exercise that is widely recommended for injury prevention. Among the benefits of stretching are an increased flexibility, enhanced muscular coordination, stress relief, improved range of motion and an improved posture. Previous studies have shown stretching training to increase arterial compliance and acutely increase sympathetic nerve activity. In addition, low flexibility levels have been found to be associated with arterial stiffness. Given that stretching of skeletal muscle causes an increase in sympathetic nerve activity; repetitive stimulation of sympathetic activity induced by habitual stretching, might chronically reduce resting sympathetic activity. The reduction in sympathetic activity might result in a decrease of arterial stiffness and blood pressure.

The investigators hypothesis is that 8 weeks of stretching training would reduce arterial stiffness, blood pressure and sympathetic activity in obese women. The investigators also hypothesize that the improved arterial function with stretching would be associated with increases in flexibility levels.

DETAILED DESCRIPTION:
The purpose of this study is to examine the effects of 8 weeks of stretching training on blood pressure,arterial stiffness, wave reflection, endothelial function and cardiovascular autonomic control. The specific aim of the study is:

- To evaluate the effects of 8 weeks of ST on arterial function and aortic hemodynamics by assessing arterial stiffness (aortic, systemic, and leg), aortic blood pressure and wave reflection, and autonomic function (heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and baroreflex sensitivity)

ELIGIBILITY:
Inclusion Criteria:

* 50-65 years old
* Blood pressure between 121/81 and 159/99 mmHg
* Body mass index of 25-39.9
* Sedentary or low active (less than 2 hr per wk)

Exclusion Criteria:

* Younger than 50 or older than 65 years of age
* Body mass index lower than 25, or 40 or higher
* Physically active or competitively active
* Smoker
* Systolic blood pressure higher than 160 mmHg
* Use of hormone replacement therapy of less than 1 yr
* Use of calcium channel blocker or beta blockers
* Type 1 diabetes
* Type 2 diabetes
* Known cardiovascular disease

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks
  Non-invasive measures of brachial and aortic blood pressure

SECONDARY OUTCOMES:
Arterial Stiffness | 8 weeks
  Using pulse wave velocity of the aorta, systemic, and legs

OTHER OUTCOMES:
Autonomic Function | 8 weeks
  Heart rate variability, vascular sympathetic activity [low-frequency power of systolic BP variability], and spontaneous baroreflex sensitivity will be assessed from electrocardiogram and beat-by-beat digital blood pressure
Pressure Wave Reflection | 8 weeks
  Using the augmentation index from radial tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, M.D., Ph.D, Study Director — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States